CLINICAL TRIAL: NCT05264376
Title: Evaluating an Eating Disorder Prevention Program for Young Women With Type 1 Diabetes
Brief Title: Eating Disorder Prevention Program for Women With T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Eric Stice, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 63675; P30DK116074 (NIH)
Record Dates: First submitted 2022-02-17; First posted 2022-03-03 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Eating Disorders; Type 1 Diabetes
MeSH Terms: conditions — Feeding and Eating Disorders; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: The Diabetes Body Project and educational control are both designed to last six weeks, for one hour each week. They both focus on diabetes-specific health issues as well as generic issues with thin-idealization.
Who Masked: Investigator
Masking Description: The research assistant conducting the diagnostic interviews after the end of the prevention program and at 3-month follow-up won't know whether the participant was in the Diabetes Body Project or the educational control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Body Project (Experimental)
  Interventions: Behavioral: Diabetes Body Project
- Educational Control Group (Active Comparator)
  Interventions: Behavioral: Educational Control

INTERVENTIONS:
Behavioral: Diabetes Body Project — The Diabetes Body Project (DBP) is an adapted version of the Body Project Prevention program designed specifically for individuals with Type 1 Diabetes. DBP consists of six weekly, one-hour long sessions. Group participants complete the exercises from the original Body Project and also new diabetes-specific content, drawn from Olmsted et al. (2002) that is delivered in a dissonance-based interactive format with Socratic questions from group leaders encourage participants to generate their own answers.
  Arms: Diabetes Body Project
Behavioral: Educational Control — We selected a T1D management/Eating disorder psychoeducational comparison condition previously tested (Olmsted et al., 2002) to control for expectancy effects and demand characteristics. To match the Diabetes Body Project, the educational lectures by Dr. Olmsted will be delivered in 6 1-hour blocks. Topics include basic information about the various EDs, complications of ED behaviors, diabetes and body image, effects of dieting on blood glucose, and the risk of complications.
  Arms: Educational Control Group

SUMMARY:
This study aims to test the effectiveness of an evidence-based eating- disorder prevention program specifically targeted for individuals with Type 1 Diabetes (T1D) compared to an educational control group. The Diabetes Body Project (DBP), is an adaptation of the Body Project which is the only eating disorder prevention program to have repeatedly produced effects when evaluated by independent researchers, produced stronger effects than credible alternative interventions, and affected objective outcomes. DBP has been adapted slightly for individuals with T1D who are at ultra-high risk for eating disorders. The study aims to test the effectiveness of the DBP of reducing body image concerns and reducing eating pathology and improving glycemic control.

ELIGIBILITY:
Inclusion Criteria:

I)female-identifying II) aged 15-30 years old III) diagnosis of T1D for at least a 6-month duration per American Diabetes Association(ADA) criteria who are taking insulin IV) have visited their diabetes care provider in the past year V) body image concerns

Exclusion Criteria:

I) not female identifying II) not in age range III) does not have a diagnosis of T1D for at least 6 months per ADA criteria who are taking insulin IV) have not visited their diabetes care provider in the past year V) do not report some level of body dissatisfaction

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, PhD, Principal Investigator — Stanford University; Korey Hood, MDPhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stice E, Gau JM, Rohde P, Shaw H. Risk factors that predict future onset of each DSM-5 eating disorder: Predictive specificity in high-risk adolescent females. J Abnorm Psychol. 2017 Jan;126(1):38-51. doi: 10.1037/abn0000219. Epub 2016 Oct 6. PMID 27709979
- [Background] Markowitz JT, Butler DA, Volkening LK, Antisdel JE, Anderson BJ, Laffel LM. Brief screening tool for disordered eating in diabetes: internal consistency and external validity in a contemporary sample of pediatric patients with type 1 diabetes. Diabetes Care. 2010 Mar;33(3):495-500. doi: 10.2337/dc09-1890. Epub 2009 Dec 23. PMID 20032278
- [Background] Fisher L, Polonsky WH, Hessler DM, Masharani U, Blumer I, Peters AL, Strycker LA, Bowyer V. Understanding the sources of diabetes distress in adults with type 1 diabetes. J Diabetes Complications. 2015 May-Jun;29(4):572-7. doi: 10.1016/j.jdiacomp.2015.01.012. Epub 2015 Feb 7. PMID 25765489
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] de Wit M, Pouwer F, Gemke RJ, Delemarre-van de Waal HA, Snoek FJ. Validation of the WHO-5 Well-Being Index in adolescents with type 1 diabetes. Diabetes Care. 2007 Aug;30(8):2003-6. doi: 10.2337/dc07-0447. Epub 2007 May 2. PMID 17475940
- [Result] Stice E, Wisting L, Desjardins CD, Hood KK, Hanes S, Rubino L, Shaw H. Evaluation of a novel eating disorder prevention program for young women with type 1 diabetes: A preliminary randomized trial. Diabetes Res Clin Pract. 2023 Dec;206:110997. doi: 10.1016/j.diabres.2023.110997. Epub 2023 Nov 10. PMID 37951479

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diabetes Body Project | Educational Control Group
Started | 30 | 25
Completed | 30 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetes Body Project | Educational Control Group | Total
Number analyzed (Participants) | 30 | 25 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 27 | 21 | 48
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 55
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 28 | 22 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 25 | 18 | 43
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 25 | 55
Thin-Ideal Internalization [Mean (Standard Deviation); unit: score on a scale] — Assessed with the 8-item Ideal-Body Stereotype Scale-Revised (Stice et al., 2017) which measures pursuit of the thin ideal. Each item is scored on a scale of 1 = strongly disagree to 5 = strongly agree. Item scores were averaged to create an overall score (1 to 5). Higher scores indicate greater belief in the thin-deal.
  score on a scale | 3.48 (.52) | 3.22 (.77) | 3.36 (0.65)
Body Dissatisfaction (BS) [Mean (Standard Deviation); unit: score on a scale] — Assessed with the 10-item Body Dissatisfaction Scale which assesses dissatisfaction with various body parts. Each item is scored on a scale of 1 = extremely dissatisfied to 6 = extremely satisfied. Item scores were averaged to create an overall score (1 to 6). Lower scores indicate greater body dissatisfaction.
  score on a scale | 3.66 (.61) | 3.46 (.83) | 3.57 (0.71)
Negative Affect [Mean (Standard Deviation); unit: score on a scale] — Negative affect will be assessed with the sadness, guilt, and fear/anxiety subscales (totaling 20 items) from the Positive Affect and Negative Affect Scale-Revised. Each item is scored on a scale of 1 = Not at All to 5 = Extremely. Item scores were averaged to create an overall score (1 to 5) Higher scores indicate greater negative affect.
  score on a scale | 2.15 (.73) | 2.38 (.89) | 2.25 (0.81)
Eating Disorder Symptoms [Mean (Standard Deviation); unit: composite score] — Eating Disorder Symptoms: Scores range from 0 to over 100 for the most severe cases. Higher scores indicate higher levels of eating disorder symptoms. Items assessing symptoms in the past month were summed to form a composite.
  composite score | 12.83 (8.65) | 16 (18.12) | 14.27 (13.73)
Diabetes eating pathology [Mean (Standard Deviation); unit: score on a scale] — Assessed with the 16-item Diabetes Eating Problem Survey-Revised. Each item is assessed on a scale of 0 = Never to 5= Always. Item scores were averaged to create an overall score (0 to 5). Higher scores indicate greater eating pathology specific to individuals with Type 1 Diabetes such as purposefully not taking enough insulin.
  score on a scale | 1.34 (.65) | 1.43 (.81) | 1.38 (0.72)
Diabetes Distress [Mean (Standard Deviation); unit: score on a scale] — Assessed with the 28-item Type 1 Diabetes Distress Scale which measures distress related to diabetes. Each item is assessed on a scale of 1 = Not a Problem to 6 = A Very Serious Problem. Item scores were averaged to create an overall score (1 to 6). High scores indicate greater distress that are related to living with Type 1 Diabetes.
  score on a scale | 2.44 (.82) | 2.44 (1.01) | 2.44 (0.9)
Quality of Life [Mean (Standard Deviation); unit: score on a scale] — Assessed with the 5-item World Health Organization Well-Being Index that measures health related quality of life. Each item is scored on a scale of 0 = At no Time to 5 = All of the Time. Item scores were averaged to create an overall score (0 to 5). Higher scores indicate greater well-being.
  score on a scale | 2.33 (.99) | 2.07 (.99) | 2.21 (0.99)
Percentage of Time With Blood Sugar in Range [Mean (Standard Deviation); unit: percentage of time] — Participants wore a continuous-glucose monitor for 14 days as well as self-reported A1c levels. The percentage of time that participants had blood sugar in range (70 to 180 mg/dL) is reported.
  percentage of time | .63 (.21) | .62 (.19) | 0.63 (0.20)
Education [Count of Participants; unit: Participants]
  Grade School | 0 | 1 | 1
  Some High School | 3 | 1 | 4
  High School Degree/Equivalent | 1 | 4 | 5
  Some College, no Degree | 4 | 7 | 11
  Associate's Degree | 2 | 1 | 3
  Bachelor's Degree | 14 | 7 | 21
  Master's Degree | 4 | 3 | 7
  Ph.D. or Higher | 2 | 0 | 2
  Did Not Disclose | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time With Blood Sugar in Range as a Measure of Glycemic Control
Description: Participants wore a continuous-glucose monitor for 14 days as well as self-reported A1c levels. The percentage of time that participants had blood sugar in range (70 to 180 mg/dL) is reported.
Time Frame: Three months following the 6-week intervention period
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Diabetes Body Project | Educational Control Group
Number analyzed (Participants) | 30 | 25
percentage of time | 0.61 (0.20) | 0.63 (0.21)

2. Primary Outcome: Eating Disorder Symptoms
Description: Participants completed a diagnostic interview using the semi-structured Eating Disorder Diagnostic Interview (EDDI) was used to assess eating disorder symptoms, including frequency of binge eating, vomiting, laxative/diuretic use, fasting, and excessive exercise, as well as degree of overvaluation of weight/shape, feeling fat, and fear of weight gain. Participants were also asked about distress regarding binge eating, rapid eating, eating until uncomfortably full, eating large quantities of food when not hungry, eating alone because of embarrassment, and feeling disgusted, depressed, or guilty after binge eating. The research assistant administering the interview was blinded to the person's condition. Scores range from 0 to over 100 for the most severe cases. Higher scores indicate higher levels of eating disorder symptoms. Items assessing symptoms in the past month were summed to form a composite.
Time Frame: Assessed at week 6 (post-intervention) and three months following the 6-week intervention period
Measure: Mean (Standard Deviation); unit: composite score
Arm/Group | Diabetes Body Project | Educational Control Group
Number analyzed (Participants) | 30 | 25
composite score
  Post-Test (week 6) | 6.50 (8.10) | 11.87 (12.42)
  3-Month Post-Test Follow Up | 5.82 (7.14) | 12.30 (14.00)

3. Primary Outcome: Body Dissatisfaction (BS)
Description: Assessed with the 10-item Body Dissatisfaction Scale which assesses dissatisfaction with various body parts. Each item is scored on a scale of 1 = extremely dissatisfied to 6 = extremely satisfied. Item scores were averaged to create an overall score (1 to 6). Lower scores indicate greater body dissatisfaction.
Time Frame: Week 6 (post-intervention) and three months following the 6-week intervention period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Body Project | Educational Control Group
Number analyzed (Participants) | 30 | 25
score on a scale
  Post-Test (week 6) | 2.98 (0.56) | 3.46 (0.50)
  3-Month Post-Test Follow Up | 3.09 (0.71) | 3.29 (0.70)

4. Primary Outcome: Thin Ideal Internalization
Description: Assessed with the 8-item Ideal-Body Stereotype Scale-Revised which measures pursuit of the thin ideal. Each item is scored on a scale of 1 = strongly disagree to 5 = strongly agree. Item scores were averaged to create an overall score (1 to 5). Higher scores indicate greater belief in the thin-deal.
Time Frame: Week 6 (post-intervention) and three months following the 6-week intervention period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Body Project | Educational Control Group
Number analyzed (Participants) | 30 | 25
score on a scale
  Post-Test (week 6) | 2.92 (0.75) | 3.15 (0.66)
  3-Month Post-Test Follow-Up | 3.12 (0.71) | 3.10 (0.65)

5. Primary Outcome: Diabetes-Specific Eating Pathology
Description: Assessed with the 16-item Diabetes Eating Problem Survey-Revised. Each item is assessed on a scale of 0 = Never to 5= Always. Item scores were averaged to create an overall score (0 to 5). Higher scores indicate greater eating pathology specific to individuals with Type 1 Diabetes such as purposefully not taking enough insulin.
Time Frame: Week 6 (post-intervention) and three months following the 6-week intervention period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Body Project | Educational Control Group
Number analyzed (Participants) | 30 | 25
score on a scale
  Post-Test (week 6) | 0.64 (0.39) | 1.02 (0.44)
  3-Month Post-Test Follow Up | 0.70 (0.48) | 1.06 (0.69)

6. Primary Outcome: Diabetes-Specific Distress
Description: Assessed with the 28-item Type 1 Diabetes Distress Scale which measures distress related to diabetes. Each item is assessed on a scale of 1 = Not a Problem to 6 = A Very Serious Problem. Item scores were averaged to create an overall score (1 to 6). High scores indicate greater distress that are related to living with Type 1 Diabetes.
Time Frame: Week 6 (post-intervention) and three months following the 6-week intervention period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Body Project | Educational Control Group
Number analyzed (Participants) | 30 | 25
score on a scale
  Post-Test (week 6) | 1.81 (0.88) | 2.08 (0.82)
  3-Month Post-Test Follow Up | 1.92 (0.96) | 2.18 (1.22)

7. Primary Outcome: Negative Affect
Description: Negative affect will be assessed with the sadness, guilt, and fear/anxiety subscales (totaling 20 items) from the Positive Affect and Negative Affect Scale-Revised. Each item is scored on a scale of 1 = Not at All to 5 = Extremely. Item scores were averaged to create an overall score (1 to 5) Higher scores indicate greater negative affect.
Time Frame: Week 6 (post-intervention) and three months following the 6-week intervention period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Body Project | Educational Control Group
Number analyzed (Participants) | 30 | 25
score on a scale
  Post Test (week 6) | 1.79 (0.77) | 2.01 (0.64)
  3-Month Post Test Follow Up | 1.95 (0.79) | 2.34 (1.09)

8. Primary Outcome: Quality of Life (Well-Being)
Description: Assessed with the 5-item World Health Organization Well-Being Index that measures health related quality of life. Each item is scored on a scale of 0 = At no Time to 5 = All of the Time. Item scores were averaged to create an overall score (0 to 5). Higher scores indicate greater well-being.
Time Frame: Week 6 (post-intervention) and three months following the 6-week intervention period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Body Project | Educational Control Group
Number analyzed (Participants) | 30 | 25
score on a scale
  Post-Test (week 6) | 2.94 (0.91) | 2.55 (0.88)
  3-Month Post-Test Follow Up | 2.75 (0.99) | 2.17 (0.93)

ADVERSE EVENTS:
Time Frame: 6-week intervention period plus 3-month follow-up period
Arm/Group | Diabetes Body Project | Educational Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/25
Other Adverse Events (participants affected / at risk) | 0/30 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/76/NCT05264376/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/76/NCT05264376/SAP_001.pdf